CLINICAL TRIAL: NCT00966914
Title: Randomized, Multicenter, Double-blind, Phase 3 Trial of Tavocept Versus Placebo in Patients With Newly Diagnosed or Relapsed Advanced Primary Adenocarcinoma of the Lung Treated With Docetaxel or Paclitaxel Plus Cisplatin
Brief Title: Phase 3 Study of Tavocept Versus Placebo in Patients With Newly Diagnosed or Relapsed Advanced Primary Adenocarcinoma of the Lung Treated With Docetaxel or Paclitaxel Plus Cisplatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioNumerik Pharmaceuticals, Inc. (Industry)
Collaborators: Lantern Pharma Inc. became Sponsor of Tavocept (BNP7787) IND 051014 as of March 26, 2019. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMS32212R
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Paclitaxel; 2,2'-dithiodiethanesulfonic acid; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo in combination with cisplatin and either paclitaxel or docetaxel
  Interventions: Drug: Placebo in combination with cisplatin and docetaxel or paclitaxel
- Tavocept (BNP7787) (Active Comparator): Tavocept (BNP7787) in combination with cisplatin and either docetaxel or paclitaxel
  Interventions: Drug: Tavocept(BNP7787) in combination with cisplatin and either docetaxel or paclitaxel

INTERVENTIONS:
Drug: Tavocept(BNP7787) in combination with cisplatin and either docetaxel or paclitaxel — Paclitaxel 200 mg/m2 IV or Docetaxel 75mg/m2 IV every 3 weeks plus Cisplatin 80 mg/m2 IV every 3weeks plus Tavocept(BNP7787) 18.4gm/m2 IV every 3 weeks
  Other Names: BNP7787
  Arms: Tavocept (BNP7787)
Drug: Placebo in combination with cisplatin and docetaxel or paclitaxel — Paclitaxel 200 mg/m2 IV or Docetaxel 75mg/m2 IV every 3 weeks plus Cisplatin 80 mg/m2 IV every 3weeks plus Placebo IV every 3 weeks
  Arms: Placebo

SUMMARY:
Tavocept is an investigational drug that is being developed to see if it can increase the survival of patients who are being treated with chemotherapy as well as to see if it can prevent or reduce side effects of chemotherapy. This research study is aimed at trying to find out if people with advanced adenocarcinoma of the lung who are treated with a standard combination of chemotherapy drugs will live longer if they are also treated with an investigational drug called "Tavocept." Another objective of this research study is to find out whether or not Tavocept helps to prevent or reduce side-effects like kidney damage, anemia, and nausea and vomiting that can occur with these drug combinations. The drug combinations that will be used in this research study will include either paclitaxel and cisplatin, or docetaxel and cisplatin. These drug combinations are approved to be used to treat people with advanced NSCLC. Every patient on this research study will be treated with standard chemotherapy for primary NSCLC in the form of either docetaxel or paclitaxel (these will be recommended by your research study doctor), which will be given in combination with cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histopathological diagnosis of inoperable advanced primary adenocarcinoma (including bronchioalveolar cell carcinoma) of the lung
* No prior systemic treatment for non-small cell lung cancer including chemotherapy, immunotherapy, hormonal therapy, targeted therapies or investigational drugs

Exclusion Criteria:

* Small cell, squamous cell, large cell or undifferentiated or any form of mixed (eg, small cell and adenocarcinoma or squamous and adenocarcinoma) histopathological or cytological diagnosis of primary lung cancer
* Adenocarcinoma arising from primary sites other than the lung
* Patients without documented Stage 4 disease (in accordance with AJCC TMM Staging System 7th edition)
* Patients with unstable CNS mets within 21 days before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival | throughout study

SECONDARY OUTCOMES:
Progression Free Survival | Every 2 cycles during study treatment then every 6-8 weeks after going off study for up to 6 months, or until progression or initiation of further treatment
Incidence of 30% or greater decrease in the calculated creatinine clearance relatively to baseline | throughout the study
Incidence of NCI-CTCAE grade 2,3, or 4 anemia | throughout the study
Proportion of patients having no impact of chemotherapy-induced emesis on daily life | throughout the study

CONTACTS AND LOCATIONS:
Locations (40):
- United States (4):
  - Birmingham, Alabama
  - Columbia, Missouri
  - Philadelphia, Pennsylvania
  - Germantown, Tennessee
- Bulgaria (4):
  - Gabrovo
  - Plovidv
  - Sofia
  - Veliko Tarnovo
- Poland (4):
  - Elblag
  - Szczecin
  - Torun
  - Warsaw
- Romania (5):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Timișoara
- Russia (15):
  - Arkangelsk
  - Chelyabinsk
  - Krasnodar
  - Krasnodar Krai
  - Kursk
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Stavropol
  - Stavropol Krai
  - Tambov
  - Voronezh
  - Yaroslavl
  - Yekaterinburg
- Ukraine (8):
  - Chernihiv
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kherson
  - Sumy
  - Uzhhorod
  - Zaporiahya